CLINICAL TRIAL: NCT07358624
Title: Patient Satisfaction and Postoperative Pain After Diagnostic Hysteroscopy: A Randomized Controlled Study Comparing Spinal and General Anesthesia
Brief Title: Patient Satisfaction and Postoperative Pain After Diagnostic Hysteroscopy: Spinal Versus General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Charles Nicolle (Other)
Responsible Party: Principal Investigator, jebri alia, Head of anesthesia and intensive care departement, Hopital Charles Nicolle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Charles Nicolle Hospital
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hysteroscopy; Patient Satisfaction; Postoperative Pain
Keywords: Diagnostic hysteroscopy; postopertive pain; patient satisfaction; anesthesia complications
MeSH Terms: conditions — Patient Satisfaction; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: GA Group: patients undergoing diagnostic hysteroscopy under general anesthesia with an I-gel supraglottic airway.
  SA Group: patients undergoing diagnostic hysteroscopy under spinal anesthesia
Who Masked: Investigator
Masking Description: patients are randomly divided into two equal groups by an investigator not directly linked to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group GA: General anesthesia (Active Comparator): Group GA: patients undergoing diagnostic hysteroscopy under general anesthesia with an I-gel supraglottic airway and post operative pain scores and patient satisfaction evaluation
  Interventions: Procedure: Group GA: post operative pain scores and patient satisfaction evaluations
- Group SA: Spinal anesthesia (Active Comparator): Group SA: patients undergoing diagnostic hysteroscopy under spinal anesthesia and post operative pain scores and patient satisfaction evaluations
  Interventions: Procedure: Group GA: post operative pain scores and patient satisfaction evaluations

INTERVENTIONS:
Procedure: Group GA: post operative pain scores and patient satisfaction evaluations — * Postoperative pain was assessed using the Numeric Rating Scale (NRS) in the post-anesthesia care unit (PACU), on postoperative day 1 and day 2.
  * Patient satisfaction with anesthesia was evaluated using the Iowa Satisfaction with Anesthesia Scale (ISAS)

SUMMARY:
Background: Diagnostic hysteroscopy is a common ambulatory gynecological procedure that may be associated with perioperative discomfort and postoperative pain. The optimal anesthetic technique for improving patient comfort while ensuring rapid recovery remains controversial. This study aimed to compare spinal anesthesia and general anesthesia with a supraglottic airway in terms of postoperative pain and patient satisfaction following diagnostic hysteroscopy.

Methods: The investigators conducted a prospective, randomized, single-blind controlled study over a four-month period in a tertiary university hospital. After obtaining informed written consent, Adult women, American Society of Anesthesiologists (ASA) physical status of I, II, or stable III, without contraindications to spinal anesthesia, known allergy to anesthetic agents, full stomach, body mass index >35 kg/m², history of migraine or communication difficulties, scheduled for diagnostic hysteroscopy were randomly assigned to receive either general anesthesia with an I-gel supraglottic airway (GA group) or spinal anesthesia (SA group). Heart rate, non invasif blood pressure and pulse oxymetry are monitored. Postoperative pain was assessed using the Numeric Rating Scale (NRS) in the post-anesthesia care unit (PACU), on postoperative day 1 and day 2. Patient satisfaction with anesthesia was evaluated using the Iowa Satisfaction with Anesthesia Scale (ISAS). Secondary outcomes included recovery time, duration of stay in the PACU, and anesthesia-related complications.

Statistical study:

Data entry and analysis were performed by SPSS software version 26.0. We used Excel 2019 software to edit the charts. We retained a significance threshold for p less than 5%.

DETAILED DESCRIPTION:
BACKGROUND : Diagnostic hysteroscopy is widely performed as an ambulatory procedure to investigate abnormal uterine bleeding, infertility, and suspected intrauterine pathology. Despite being minimally invasive, it may generate discomfort and postoperative pain, particularly during cervical dilation and uterine distension. Choosing an anesthetic technique that optimizes patient comfort while preserving rapid recovery is therefore crucial.

General anesthesia with short-acting agents and supraglottic airway devices is commonly used in the operating room because it provides predictable conditions and fast emergence; however, it may be associated with postoperative nausea and vomiting and hemodynamic instability. Spinal anesthesia provides effective analgesia and stable surgical conditions, but may result in hypotension, urinary retention, post-dural puncture headache, and occasional failure requiring conversion to general anesthesia. Current evidence comparing these techniques in diagnostic hysteroscopy remains conflicting, and patient satisfaction-an important outcome in ambulatory care-has not been consistently evaluated.

This study compared spinal anesthesia and general anesthesia with a supraglottic airway in women undergoing diagnostic hysteroscopy, focusing on postoperative pain and patient satisfaction, as well as recovery outcomes and anesthesia-related adverse events.

Methods:

Study Design and Setting This prospective, randomized, single-blind controlled study was conducted over a four-month period, from September to December 2024, in the operating rooms of the Gynecology Departments A and B of Charles Nicolle University Hospital, Tunis.

Participants Adult women (≥18 years) scheduled for diagnostic hysteroscopy were screened during the pre-anesthetic consultation.

Randomization and Blinding:

Eligible patients were randomly assigned to one of two groups: general anesthesia (GA group) or spinal anesthesia (SA group). Randomization was performed preoperatively. Patients were blinded to the anesthetic technique used, whereas the anesthesiologist was not.

Anesthetic Management:

General Anesthesia: Patients in the GA group received preoxygenation followed by intravenous induction with fentanyl (approximately 3 μg/kg) and propofol (approximately 3 mg/kg). A supraglottic airway device (I-gel®) was inserted once adequate depth of anesthesia was achieved. Mechanical ventilation was provided in volume-controlled mode with lung-protective settings. Anesthesia was maintained with a continuous propofol infusion adjusted to achieve a Ramsay sedation score of 5. Intravenous paracetamol (1 g) was administered intraoperatively for postoperative analgesia. The supraglottic airway was removed after recovery of protective airway reflexes.

Spinal Anesthesia: In the SA group, spinal anesthesia was performed under aseptic conditions at the L3-L4 or L4-L5 interspace using a 25-gauge spinal needle. After confirmation of free cerebrospinal fluid flow, a mixture of hyperbaric bupivacaine 0.5% (8 mg) and sufentanil (2.5 μg) was injected intrathecally. Oxygen was administered via nasal cannula at 2 L/min. Surgery was initiated once a sensory block level of at least T10 was achieved.

Perioperative Monitoring and Management:

Standard monitoring included non-invasive blood pressure, continuous electrocardiography, pulse oximetry, and temperature measurement and (with respiratory parameters in GA groupe). Hypotension (defined as a decrease ≥20% from baseline) was treated with intravenous ephedrine boluses, and bradycardia (HR ≤ 50 beats/min) was treated with atropine as needed. Perioperative complications were recorded.

Postoperative Management and Outcomes:

All patients were transferred to the post-anesthesia care unit (PACU). Postoperative pain was assessed using the Numeric Rating Scale (NRS) in the PACU, on postoperative day 1, and day 2. Analgesic consumption and anesthesia-related adverse events were recorded. Patient satisfaction with anesthesia was evaluated before discharge using the Iowa Satisfaction with Anesthesia Scale (ISAS). Discharge readiness from the PACU was assessed using the modified Aldrete score, and readiness for home discharge was evaluated using the Post-Anesthetic Discharge Scoring System (PADSS).

Primary outcomes : patient satisfaction and pain scores. Secondary outcomes: PACU discharge delays, home discharge delays, frequency of nausea and vomiting, headache and bladder globe.

- Statistical Analysis: Sample size calculation was based on previously published data comparing postoperative pain scores between anesthetic techniques, with a power of 80% and a significance level of 5%. Data were analyzed using IBM SPSS Statistics (version 26). Continuous variables were expressed as mean ± standard deviation and compared using Student's t-test or the Mann-Whitney U test, as appropriate. Categorical variables were expressed as frequencies and percentages and compared using the chi-square test or Fisher's exact test. Multivariate logistic regression analysis was performed to identify factors independently associated with postoperative pain and patient satisfaction. A p value ≤0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent.
* an American Society of Anesthesiologists (ASA) physical status of I, II, or stable III in
* women scheduled for diagnostic hysteroscopy

Exclusion Criteria:

* operative hysteroscopy.
* contraindications to spinal anesthesia.
* known allergy to anesthetic agents.
* full stomach.
* body mass index >35 kg/m².
* history of migraine.
* communication difficulties

Patients were excluded from the final analysis in case of:

* spinal anesthesia failure requiring conversion to general anesthesia.
* failure of ventilation with a supraglottic airway requiring tracheal intubation.
* conversion to laparotomy.
* prolonged hospitalization for non-anesthesia-related complications.
* loss to follow-up after discharge.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Pain scores evaluation | Pain score was evaluated up to the second post operative day
  Numeric Rating Scale (minimum =1 maximum =10; 1-3:mild pain; 4-7:moderate pain; 8-10:severe pain) in the post-anesthesia care unit (PACU), on postoperative day 1 and day 2 was evaluated
patient satisfaction | Iowa Satisfaction with Anesthesia Scale is evaluated in the post operative first hour (11 statements; usually 6 choices from "strongly disagree" to "strongly agree"were evaluated;
  Patient satisfaction with anesthesia was evaluated using the Iowa Satisfaction with Anesthesia Scale (ISAS)

SECONDARY OUTCOMES:
anesthesia complications | anesthesia complications was recorded in the post operative first day
  frequency of post operative nausea and vomiting , headache and bladder globe
duration of stay in the PACU | duration of stay in the PACU was evaluated in the postopertive second hour
  PACU discharge was determined by modified Aldrete score (Minimum score = 0; maximum score = 10; discharge is permitted if score ≥ 9)
recovery time | ome discharge delays was evaluated in the postoperative first four hours
  home discharge delays

CONTACTS AND LOCATIONS:
Overall Officials: Alia Jebri, MD, Study Director — Charles Nicolle Hospital Tunis
Locations (1):
- Charles Nicolle hospital Tunis, Bab Saadoun, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nzau-Ngoma E, Odimba M, Kusuman A, Mboloko E. Office hysteroscopy: findings in patients attending a clinic in Kinshasa. The international society of endoscopic gynecology. 2022;
- [Background] Samy A, Nabil H, Abdelhakim AM, Mahy ME, Abdel-Latif AA, Metwally AA. Pain management during diagnostic office hysteroscopy in postmenopausal women: a randomized study. Climacteric. 2020 Aug;23(4):397-403. doi: 10.1080/13697137.2020.1742685. Epub 2020 Apr 17. PMID 32299254
- [Background] Manouchehrian N, Pilehvari S, Rahimi-Bashar F, Esna-Ashari F, Mohammadi S. Comparison of the effects of spinal anesthesia, paracervical block and general anesthesia on pain, nausea and vomiting, and analgesic requirements in diagnostic hysteroscopy: A non-randomized clinical trial. Front Med (Lausanne). 2023 Mar 1;10:1089497. doi: 10.3389/fmed.2023.1089497. eCollection 2023. PMID 36936226
- [Background] The Use of Hysteroscopy for the Diagnosis and Treatment of Intrauterine Pathology: ACOG Committee Opinion, Number 800. Obstet Gynecol. 2020 Mar;135(3):e138-e148. doi: 10.1097/AOG.0000000000003712. PMID 32080054
- [Background] Stefanescu A, Marinescu B. Diagnostic hysteroscopy - a retrospective study of 1545 cases. Maedica (Bucur). 2012 Dec;7(4):309-14. PMID 23483793
- [Background] Centini G, Troia L, Lazzeri L, Petraglia F, Luisi S. Modern operative hysteroscopy. Minerva Ginecol. 2016 Apr;68(2):126-32. Epub 2016 Mar 1. PMID 26930389